CLINICAL TRIAL: NCT02502175
Title: Comparing Opium Tincture (OT) and Methadone for Medication-assisted Treatment of Opioid Use Disorder: A Randomized Double-blind Controlled Clinical Trial
Brief Title: Comparing Opium Tincture (OT) With Methadone for Medication-assisted Treatment of Opioid Use Disorder
Acronym: OT-RCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Tehran University of Medical Sciences (Other); Iran National Science Foundation (Unknown); AJA University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Michael Krausz, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H15-00220
Record Dates: First submitted 2015-07-13; First posted 2015-07-20 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Opioid Dependence
Keywords: Opium tincture; opium; methadone; opioid dependence; opiate dependence; clinical trial; Iran
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Opium; Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opium (Experimental): patient-centered flexible dosing in line with the national protocol published by Iranian Ministry of Health for maintenance treatment of opioid dependent population
  Interventions: Drug: opium
- methadone (Active Comparator): patient-centered flexible dosing in line with the national protocol published by Iranian Ministry of Health for maintenance treatment of opioid dependent population
  Interventions: Drug: methadone

INTERVENTIONS:
Drug: opium — Opium tincture (10mg/ml), manufactured by Daroupakhsh.co, Tehran, Iran.
  Other Names: tincture of opium; laudanum; Opium tincture
  Arms: Opium
Drug: methadone — Methadone (5mg/ml), manufactured by Daroupakhsh.co, Tehran, Iran.
  Arms: methadone

SUMMARY:
Patients with opioid use disorder seeking medication-assisted treatment will be recruited. Each participant will be allocated to one of the two study groups with the equal chance of receiving either opium tincture (OT) or methadone. Participants, clinical and research staff will not be aware of the medication that each patient receives. This study aims to test whether OT is as equally effective as methadone at retaining participants with opioid use disorder in medication-assisted treatment.

DETAILED DESCRIPTION:
Purpose:

To compare the efficacy and safety of opium tincture (OT) with methadone syrup for medication-assisted treatment of individuals with opioid use disorder.

Justification:

Currently, methadone is the gold standard for medication-assisted treatment of opioid use disorder. Opium tincture could be a potential alternative treatment for this condition, and a promising solution to address the following issues:

1. Alternative treatment option As no single treatment is effective for all individuals with opioid use disorder, sufficiently diverse treatment options should be available. Currently, treatment options for opioid use disorder are not always effective.
2. Avoidance of overdose with methadone:

   The long-acting nature of methadone, its narrow therapeutic window, its high potency and associated lack of standard conversion ratio from and to other drugs, could result in fatal overdose. In contrast, OT has a shorter half-life and lower potency compared to methadone, which can account for a lower incidence of fatal overdose, especially in patients at higher risk of overdose with currently prescribed medications. Thus, OT could be an added treatment option to currently available treatments such as Buprenorphine/ Naloxone for medication-assisted treatment of patients with higher risk of overdose.
3. Prolonged QT syndrome of methadone:

   Medication-assisted treatment with methadone can cause serious, potentially fatal adverse effects on the cardiac electrical conduction system leading to a prolonged QT interval and predisposing patients to arrhythmias. As such, cardiac conduction co-morbidity is a (relative) contraindication for the use of methadone as a medication-assisted treatment. Thus, OT could be an added treatment option to current available treatments such as buprenorphine or levomethadone for medication-assisted treatment of patients with cardiac conduction defects.
4. Opium dependence as the dominant pattern of substance use To date, studies on medication-assisted treatment of opioid use disorder have mostly been carried out on populations in which heroin is the predominant substance of use and there is comparatively fewer data on patients with opium use disorder. Opium tincture could be the treatment of choice in geographic areas with higher prevalence of dependence on opium as the predominant pattern of substance use, such as Iran and some other Asian countries.
5. Traditional medicine and cultural acceptance: Being a traditional herbal remedy for pain, OT appears to be a more culturally acceptable alternative to methadone in some parts of Southeast Asia.
6. Cost-effectiveness: Possible cost effectiveness of OT for treatment of opioid use disorder can make it a potential treatment of choice if its efficacy and safety profile could be demonstrated through this RCT.

Research methods:

1. Recruitment strategy: Following methods will be used to recruit participants: 1) Brochures and flyers will be distributed in community outreach, general and mental hospitals, NGO-run communities, colleges and universities, drop-in centers and specialized clinics for treatment of participants with HIV and hepatitis C 2) Posters (same content as a brochures and flyers) of the study will be stuck in the billboard of bus/subway, local stores, hospitals, NGO-run communities, colleges and universities, as well as any specialized health-care center for psychiatry or addiction treatments 3) there are NGO-run communities for treating patients with opioid use disorder in Sari, Isfahan, and Shiraz. Investigators will use the initial contact letter to recruit from new patients attending these communities for receiving treatment.
2. Randomization and blinding: Randomized to methadone or OT treatment arms will be carried out in a 1:1 allocation ratio using stratified randomization block technique with block sizes of 2. Age and gender distribution of the population with opioid-dependence in Iran is the basis for stratification on sex (F/M ratio = 1/9) and age (younger than 30/ 30-49/ 50 and older ~ 1: 2: 2). The investigators, treatment team (except pharmacist), assessors, and patients will only be aware of the randomization code for each participant, but not the treatment allocation label or randomization tables. Methadone syrup is made similar to OT in terms of smell, color, and taste using an essence.
3. Sample size: The sample size was calculated using a fixed margin (95%-95%) approach based on the FDA guidelines for non-inferiority clinical trials (Food and Drug Administration, 2016). For the active control effect, a pooled 95% CI for retention ratio of methadone to placebo of 4.44 [3.26, 6.04] was considered (Mattick et al., 2009). The lower bound i.e., 3.26 was considered as M1, with calculated treatment effect of 2.26. M2 equal to 1.25 (11% of M1) was chosen as a conservative non-inferiority margin. Retention rate for participants in medication-assisted treatment with methadone was assumed to be 77.7% at 3 months based on a comprehensive systematic review (Feelemyer et al., 2014). Based on formula by Zhong, 2009, and assuming a power of 90% and Type I error set at 5%, the total sample size was initially calculated to be 240 participants, 120 in each group. Due to financial constraints, recruitment was set to stop at 200 given that it still provides a power more than 80% (a sample size of 174 provides a power of 80%).
4. Statistical analysis plan: Retention in treatment will be compared between two groups using confidence interval procedure. Secondary outcomes will be compared between two groups using appropriate regression methods.

ELIGIBILITY:
Inclusion Criteria:

* Opioid dependence as confirmed by DSM V diagnostic criteria
* Willingness and ability to adhere to study protocol and follow-up schedule as determined through the pre-randomization period
* Provide written informed consent.
* Females of childbearing capacity must agree to use an acceptable method of birth control approved by the study investigator throughout the study.

Exclusion Criteria:

* Active participant in another treatment program for opioid dependence within 14 days before inclusion in the study
* Severe hepatic impairment (decompensated liver disease), a contraindication for methadone and its potential to precipitate hepatic encephalopathy.
* Hypersensitivity to methadone syrup or other ingredients in the formulation
* Pregnancy
* Severe chronic respiratory disease
* Head injury and raised intracranial pressure: Respiratory depressant effects (with CO2 retention and secondary elevation of CSF pressure) may be markedly exaggerated in the presence of head injury, or a preexisting increase in intracranial pressure. May produce effects that obscure the clinical course in participants with head injuries.
* Biliary tract disease: may cause constriction of sphincter of Oddi.
* Monoamine oxidase inhibitors use within 14 days of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
Retention in treatment | three months
  percent of participants retained in the treatment

SECONDARY OUTCOMES:
Craving | Day 1-3/ Twice daily | Day 4-14/ Once daily | Day 15-28/ Three times a week | Day 29-84/ Once weekly
  Visual analogue scale (0-10 scale)
Withdrawal symptoms | Day 1-3/ Twice daily | Day 4-14/ Once daily | Day 15-28/ Three times a week | Day 29-84/ Once weekly
  Subjective Opioid Withdrawal Scale (SOWS) Questionnaire
Physical health | Baseline, month 1, 2 and 3
  Opiate Treatment Index (OTI)-Health section Questionnaire
Mental health | Baseline, month 1, 2 and 3
  Symptom Checklist-90-Revised (SCL90-R) Questionnaire
Cognitive function | Baseline, month 1, 2 and 3
  Montreal Cognitive Assessment (MOCA) Questionnaire
Severity of substance use problem | Baseline, month 1, 2 and 3
  Addiction Severity Index-5th (ASI-5th) Questionnaire
Quality of life score from World Health Organization Quality of Life-BREF Questionnaire | Baseline, month 1, 2 and 3
  World Health Organization Quality of Life-BREF (WHOQoL-BREF) Questionnaire
Client Satisfaction | month 3
  Treatment Perception Questionnaire (TPQ)
Abstinence | Baseline, month 1, 2 and 3
  Use of illicit opioids: Self-report / Use of amphetamines, methamphetamines, benzodiazepines: Self-report AND urine toxicology
Adverse events | Day 1-3/ Twice daily | Day 4-14/ Once daily | Day 15-28/ Three times a week | Day 29-84/ Once weekly
  Spontaneous reports AND checklist included in the Case Report Form (CRF), physical examination and lab data
Cost-effectiveness | three months
  Cost per Quality-adjusted life-month (QALM) and Quality-adjusted life-year (QALY) is calculated using Substance Abuse Services Cost Analysis Program (SASCAP).

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Kausz, MD, PhD, Principal Investigator — University of British Columbia; Shahin Akhondzadeh, PhD, Principal Investigator — Tehran University of Medical Sciences
Locations (4):
- Iran (4):
  - Dodange Substance use disorder treatment center, Moḩammadābād, Mazandaran
  - Kian substance use treatment center, Sari, Mazandaran
  - Tavalodi Digar, Isfahan
  - Rooz-e-No substance use treatment center, Shiraz

REFERENCES:
- [Derived] Nikoo M, Kianpoor K, Nikoo N, Javidanbardan S, Kazemi A, Choi F, Vogel M, Gholami A, Tavakoli S, Wong JSH, Moazen-Zadeh E, Givaki R, Jazani M, Mohammadian F, Moghaddam NM, Schutz C, Jang K, Akhondzadeh S, Krausz M. Opium tincture versus methadone for opioid agonist treatment: a randomized controlled trial. Addiction. 2023 Feb;118(2):284-294. doi: 10.1111/add.16030. Epub 2022 Sep 7. PMID 35971297
- [Derived] Nikoo M, Moazen-Zadeh E, Nikoo N, Javidanbardan S, Kazemi A, Choi F, Vogel M, Gholami A, Tavakoli S, Givaki R, Jazani M, Mohammadian F, Markazi Moghaddam N, Goudarzi N, Schutz C, Jang K, Akhondzadeh S, Krausz M. Comparing opium tincture and methadone for medication-assisted treatment of patients with opioid use disorder: Protocol for a multicenter parallel group noninferiority double-blind randomized controlled trial. Int J Methods Psychiatr Res. 2019 Mar;28(1):e1768. doi: 10.1002/mpr.1768. Epub 2019 Feb 4. PMID 30714249